CLINICAL TRIAL: NCT03364920
Title: Serum Maresin-1 Level Predicts the Disease Severity and Clinical Outcomes of Severe Acute Pancreatitis Patients
Brief Title: Serum Maresin-1 Predicts the Severity of Severe Acute Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Weiqin Li (Other)
Responsible Party: Sponsor-Investigator, Weiqin Li, Doctor, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Other Study IDs: SMPSSAP
Record Dates: First submitted 2017-11-23; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Pancreatitis, Acute
Keywords: Maresin-1; SAP; IPN; MODS; Mortality
MeSH Terms: conditions — Pancreatitis; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal level of serum maresin-1
- abnormal level of serum maresin-1

SUMMARY:
This is a retrospective study about serum Maresin-1 level in different severe acute pancreatitis patients. The investigators want to study the correlation between the level of serum Maresin-1 and the severity of SAP, of course the clinical outcomes. The investigators want to find some biomarkers and strategy target drugs of severe acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Severe Acute Pancreatitis
* Biliary pancreatitis
* 7 days of the onset

Exclusion Criteria:

* Surgical patients
* Serious diseases and infection
* Alcoholic pancreatitis
* Hypertriglyceridemia pancreatitis
* Disorder of Glucolipide Metabolism：diabetes mellitus, hypertriglyceridemia, BMI>30

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes severe acute pancreatitis between 18ys and 75ys.Patients with disorder of glucolipide metabolism will be excluded. Alcoholic pancreatitis and HTG-AP patients will be also excluded. Patients will be divided into 2 groups according to their level of serum maresin-1.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
mortality | up to 28 days
  The level of serum maresin-1 predicts the severity of severe acute pancreatitis

SECONDARY OUTCOMES:
The incidence of MODS | through study completion, an average of 1 year
  The level of serum maresin-1 predicts the severity of severe acute pancreatitis
The incidence of IPN | through study completion, an average of 1 year
  The level of serum maresin-1 predicts the severity of severe acute pancreatitis